CLINICAL TRIAL: NCT04596423
Title: Sief_Twist Sign a Novel View in Fetal Echocardiography
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sief el eslam Ahmed Ali, Principal Investigator, Assiut University
Other Study IDs: AUE202010
Record Dates: First submitted 2020-10-15; First posted 2020-10-22 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Fetal Echocardiography

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- A: Extended fetal heart examination
  Interventions: Diagnostic Test: Fetal echocardiography
- B: Modified extended heart examination
  Interventions: Diagnostic Test: Fetal echocardiography
- C: Sief_Twist sign only examination
  Interventions: Diagnostic Test: Fetal echocardiography

INTERVENTIONS:
Diagnostic Test: Fetal echocardiography — fetal heart examination by medical ultrasound

SUMMARY:
To describe Sief_twist sign as a novel sign in fetal echocardiography as a new ,easy , time effective view in fetal heart examination .

ELIGIBILITY:
Inclusion Criteria:

1. Singleton fetus .
2. gestational age 14-37 weeks.
3. no maternal medical disorder .
4. no morbed obisity.

Exclusion Criteria:

1. evidence of fetal infection.
2. chorioamnionitis.
3. fetal anomalies.
4. abnormal fetal karyotype
5. patient withdrawal from the study and/or unavailability for follow-up.

Ages: 18 Years to 35 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — female
Study Population: observational study conducted at academic perinatal center that investigates Sief_Twest sign as novel sign in fetal heart examination in comparison with classic standard views Patients who give written consent to participate in the study undergo a uniform antenatal assessment protocol that includes basic obstetrics ultrasound examination , fetal anatomy scan & fetal echocardiography .
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2024-02-04 (Actual)

PRIMARY OUTCOMES:
obtaining clear images for fetal cardiac structures via standard views which is 4 chamber view[4CH.], left outflow tract view[LVOT.] , right outflow tract view [RVOT.], three vesseles trachea view [3VTV.] | 15 miutes
  4 chamber view that describe 4 heart chambers which are 2 atria , 2 ventricles - LVOT. view describes outflow of aorta from left ventricle in normal heart - RVOT describe outflow of pulmonary from rt. ventricle in normal heart - 3VTV describes view of aorta, pulonary and superior viena cava at upper chest

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt